CLINICAL TRIAL: NCT05642611
Title: Ice Compress: Randomized Trial of Limb Cryocompression Versus Continuous Compression Versus Low Cyclic Compression for the Prevention of Taxane-Induced Peripheral Neuropathy
Brief Title: Comparing Cooling and/or Compression Approaches of Limbs for Prevention of Chemotherapy-Induced Peripheral Neuropathy
Acronym: ICE COMPRESS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: S2205; NCI-2022-09251 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); SWOG-S2205 (Other: SWOG); SWOG-S2205 (Other: DCP); SWOG-S2205 (Other: CTEP); UG1CA189974 (NIH)
Record Dates: First submitted 2022-11-30; First posted 2022-12-08 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Malignant Solid Neoplasm
MeSH Terms: interventions — Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Cryocompression) (Experimental): Patients undergo cryocompression (cooling plus moderate and low pressure to the arms and legs) for 30-minutes pre-taxane chemotherapy infusion, during taxane chemotherapy infusion, and for 30 minutes after completion of each taxane infusion. Patients may also undergo collection of blood, serum and plasma samples during screening and on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Cryocompression Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm 2 (Continuous Compression) (Experimental): Patients undergo continuous compression (moderate, steady pressure to the arms and legs) for 30-minutes pre-taxane chemotherapy infusion, during taxane chemotherapy infusion, and for 30 minutes after completion of each taxane infusion. Patients may also undergo collection of blood, serum and plasma samples during screening and on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Pneumatic Compression Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm 3 (Low Cyclic Compression) (Active Comparator): Patients undergo low cyclic compression (low pressure that comes and goes to the arms and legs) for 30-minutes pre-taxane chemotherapy infusion, during taxane chemotherapy infusion, and for 30 minutes after completion of each taxane infusion. Patients may also undergo collection of blood, serum and plasma samples during screening and on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Pneumatic Compression Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood, plasma, and serum
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Cryocompression Therapy — Undergo cryocompression
  Arms: Arm 1 (Cryocompression)
Procedure: Pneumatic Compression Therapy — Undergo continuous compression
  Arms: Arm 2 (Continuous Compression)
Procedure: Pneumatic Compression Therapy — Undergo low cyclic compression
  Arms: Arm 3 (Low Cyclic Compression)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase III trial compares the effect of 3 study approaches in preventing chemotherapy-induced peripheral neuropathy: 1) cryocompression, 2) continuous compression, and 3) low cyclic compression. Taxane chemotherapy drugs, such as paclitaxel or docetaxel, can cause a nerve disorder called peripheral neuropathy, which can cause numbness, tingling, or pain in the arms and legs. The 3 study approaches will use a device, called the Paxman Limb Cryocompression System, made of wraps that cool and/or compress the arms and legs. This study may help researchers determine if any of the study approaches are able to prevent taxane chemotherapy from causing peripheral neuropathy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the proportion of participants who develop clinically meaningful chemotherapy induced peripheral neuropathy (CIPN) at 12 weeks, in participants treated with taxane-based chemotherapy randomized to cryocompression therapy versus continuous compression therapy versus low cyclic compression therapy.

SECONDARY OBJECTIVES:

I. To compare trajectories over time (6, 12, 24, and 52 weeks) by intervention study arm in clinically meaningful CIPN.

II. To compare mean European Organization for Research and Treatment of Cancer Chemotherapy-Induced Peripheral Neuropathy 20 (EORTC-CIPN-20) sensory neuropathy subscale scores at 12 weeks by intervention study arm.

III. To compare differences by intervention study arm at 12 weeks in changes from baseline in objective sensory and motor function tests (Neuropen, tuning fork, Timed Get Up and Go test).

IV. To compare the proportion of participants who develop clinically meaningful CIPN at 12 weeks in a sensitivity analysis with dropouts treated as failures.

V. To compare rates of adverse events related to study device at 12 weeks (including cold intolerance, skin changes, other adverse events [AEs] as assessed by Common Terminology Criteria for Adverse Events [CTCAE]) between the three interventions.

ADDITIONAL OBJECTIVES:

I. To compare the proportion of participants who develop clinically meaningful CIPN separately at weeks 6, 24, and 52.

II. To compare the proportion of participants who develop clinically meaningful CIPN at week 12 with additional covariate adjustment for age and body mass index (BMI).

III. To compare differences by intervention study arm at 12 weeks in mean EORTC CIPN-20 motor subscale score and autonomic subscale score, and in mean individual Patient-Reported Outcomes Measurement Information System (PROMIS)-29 domain (Physical Functioning, Anxiety, Depression, Fatigue, Sleep Disturbance, Social Functioning, Pain Interference, and Pain Intensity) scores.

IV. To compare trajectories over time (6, 12, 24, and 52 weeks) by intervention study arm in mean EORTC CIPN-20 sensory neuropathy subscale score, motor subscale score, and autonomic subscale score; and in mean PROMIS-29 individual domains (Physical Functioning, Anxiety, Depression, Fatigue, Sleep Disturbance, Social Functioning, Pain Interference, and Pain Intensity) scores; and in changes in objective sensory and motor function tests (Neuropen, tuning fork, Timed Get Up and Go test).

V. To evaluate the differences by intervention study arm in proportion of participants who develop clinically meaningful CIPN at 12 weeks by chemotherapy regimen.

VI. To assess the effect of the intervention in reducing CIPN occurring in the upper extremities and, separately, in the lower extremities.

VII. To explore the relationship between duration of intervention received at the prescribed level and outcome, analogous to a dose-delivered analysis in a treatment trial.

VIII. To compare rates by study arm of CTCAE Grade 2 or higher sensory and motor neuropathy at 12 weeks.

IX. To evaluate tolerability of cryocompression compared to continuous compression therapy and low cyclic compression therapy, as assessed by rate of temperature and/or pressure adjustments, interruptions, and early discontinuation of the device.

X. To determine participant satisfaction of cryocompression compared to continuous compression therapy and low cyclic compression therapy, assessed by patient questionnaire.

XI. To compare taxane dose-reductions, treatment delays/discontinuation due to CIPN, and relative taxane dose intensity and total taxane dose received, between intervention study arms.

XII. To evaluate differences of intervention effect by sex, race, and ethnicity.

XIII. To confirm pretreatment biomarkers of CIPN risk (vitamin D) and on-treatment biomarker changes indicative of CIPN severity (Neurofilament light chain, NFL) as well as additional biomarkers of interest generated in S1714 for validation.

BANKING OBJECTIVE:

I. To bank specimens for future correlative studies.

OUTLINE: Patients are randomized to 1 of 3 arms.

ARM 1: Patients undergo cryocompression (cooling plus moderate and low pressure to the arms and legs) for 30-minutes pre-taxane chemotherapy infusion, during taxane chemotherapy infusion, and for 30 minutes after completion of each taxane infusion. Patients may also undergo collection of blood, serum and plasma samples during screening and on study.

ARM 2: Patients undergo continuous compression (moderate, steady pressure to the arms and legs) for 30-minutes pre-taxane chemotherapy infusion, during taxane chemotherapy infusion, and for 30 minutes after completion of each taxane infusion. Patients may also undergo collection of blood, serum and plasma samples during screening and on study.

ARM 3: Patients undergo low cyclic compression (low pressure that comes and goes to the arms and legs) for 30-minutes pre-taxane chemotherapy infusion, during taxane chemotherapy infusion, and for 30 minutes after completion of each taxane infusion. Patients may also undergo collection of blood, serum and plasma samples during screening and on study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a diagnosis of a solid tumor malignancy.
* Participants must be planning to begin neoadjuvant or adjuvant therapy with one of the protocol-specified chemotherapy regimens below for a solid tumor malignancy within 3 calendar days after randomization.

  * Weekly paclitaxel x 12 consecutive weeks
  * Weekly paclitaxel x 12 consecutive weeks + carboplatin (weekly x 12 consecutive weeks or every 3 weeks x 4 consecutive cycles)
  * Paclitaxel + carboplatin every 3 weeks x 6 consecutive cycles without chemotherapy pause for surgery
  * Docetaxel + carboplatin every 3 weeks x 6 consecutive cycles without chemotherapy pause for surgery NOTE: For any of the protocol-specified chemotherapy regimens, concurrent targeted therapy with biologic therapy is allowed. Pembrolizumab (or other immune checkpoint inhibitors), trastuzumab and/or pertuzumab, or bevacizumab are allowed.
* Participant must be >= 18 years old.
* Participants must be offered the opportunity to participate in specimen banking. With participant consent, specimens must be collected and submitted via the Southwest Oncology Group (SWOG) Specimen Tracking System.
* Participants must be able to complete Patient-Reported Outcome (PRO) questionnaires in English or Spanish.
* Participants must 1) agree to complete PROs at all scheduled assessments, and 2) complete the baseline PRO questionnaires within 14 days prior to randomization
* Participants must be informed of the investigational nature of this study and must sign and give informed consent in accordance with institutional and federal guidelines.

For participants with impaired decision-making capabilities, legally authorized representatives may sign and give informed consent on behalf of study participants in accordance with applicable federal, local, and Central Institutional Review Board (CIRB) regulations.

Exclusion Criteria:

* Participants must not have a history of skin or limb metastases.
* Participants must not have previously received neurotoxic chemotherapy for any reason (e.g., taxanes, platinum agents, vinca alkaloids, or bortezomib).
* Participants must not have pre-existing clinical peripheral neuropathy from any cause.
* Participants must not have a history of Raynaud's phenomenon, cold agglutinin disease, cryoglobulinemia, cryofibrinogenemia, post-traumatic cold dystrophy, or peripheral arterial ischemia.
* Participants must not have any open skin wounds or ulcers of the limbs at the time of randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 777 (Estimated)
Dates: Start 2023-06-06 (Actual); Primary Completion 2030-08-01 (Estimated); Study Completion 2031-08-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence of clinically meaningful chemotherapy induced peripheral neuropathy (CIPN) (binary outcome: yes vs. no) | At the 12-week assessment after randomization
  Defined as an absolute increase of 8 or more points over baseline in the CIPN-20 sensory neuropathy subscale score. Analysis will be conducted multivariable logistic regression, adjusting for the baseline score and the stratification factor as covariates.

SECONDARY OUTCOMES:
Mean sensory neuropathy scores | At 12 weeks
  Will assess by study arm. Will examine the CIPN-20 sensory neuropathy subscale score as a continuous variable on the 0-100 scale. The differences by intervention study arm at 12 weeks in changes from baseline in objective sensory and motor function tests (Neuorpen, tuning fork, Get Up and Go test) will also be compared. Multiple linear regression analysis will be conducted, adjusting for the baseline score and the stratification factor as covariates.
Dropouts | Prior to the week 12 assessment
  Any dropouts prior to the week 12 assessment as failures. Since death is anticipated to be unrelated to the intervention assignment, deaths will be censored. Failures will be analyzed with an aggregate failure variable defined as: experience of neuropathy according to the CIPN-20 sensory neuropathy subscale score or dropout prior to week 12 (yes vs. no). Logistic regression will be used, adjusted for the stratification factor as a covariate.
Trajectories over time | 6, 12, 24, and 52 weeks
  Trajectories over time by intervention study arm in clinically meaningful CIPN will be compared. Generalized estimating equations with a logit link and robust standard errors will be used, adjusting for the baseline score and the stratification factor as covariates.
Rates of adverse events | At 12 weeks
  Rates of adverse events related to study device (including cold intolerance, skin changes, other AEs as assessed by (National Cancer Institute Common Terminology Criteria for Adverse Events [NCI-CTCAE]) between the three interventions will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa K Accordino, Principal Investigator — SWOG - Columbia University; Katherine Pennington, MD, Principal Investigator — NRG - University of Washington
Locations (29):
- United States (29):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Contra Costa Regional Medical Center, Martinez, California
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - The Valley Hospital - Luckow Pavilion, Paramus, New Jersey
  - Valley Health System Ridgewood Campus, Ridgewood, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - CaroMont Regional Medical Center, Gastonia, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Rhode Island Hospital, Providence, Rhode Island
  - McLeod Regional Medical Center, Florence, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - MGC Hematology Oncology-Union, Union, South Carolina
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - University of Washington Medical Center - Montlake, Seattle, Washington